CLINICAL TRIAL: NCT03987594
Title: Prospective Randomized Controlled Trial Comparing the Effect of Fulguration Versus Fulguration and Hydrodistension in Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Comparing the Effect of Fulguration Versus Fulguration and Hydrodistension in Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0492; 2016-12-007-001 (Other: Ewha Womans University Mokdong Hospital)
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Interstitial Cystitis; Painful Bladder Syndrome; Hydrodistension; Transurethral Fulguration
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: 1:1 allocation with Permuted block randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUF (Placebo Comparator): Subjects allocated into TUF+HD group receive bladder hydrodistension prior to transurethral fulguration of Hunner lesion
  Interventions: Procedure: Transurethral fulguration of the Hunner lesion
- TUF+HD (Experimental): Subjects allocated into TUF+HD group receive bladder hydrodistension prior to transurethral fulguration of Hunner lesion
  Interventions: Procedure: Combination treatment of bladder hydrodistension and transurethral fulguration of the Hunner lesion

INTERVENTIONS:
Procedure: Transurethral fulguration of the Hunner lesion — Hunner lesion of the bladder is fulgurated with electronic surgical device under cystoscopic inspection. For the intervention, general or spinal anesthesia is required.
  Arms: TUF
Procedure: Combination treatment of bladder hydrodistension and transurethral fulguration of the Hunner lesion — Prior to Hunner lesion fulguration, bladder hydrodistension is performed for 8 minutes at pressure of 80cmH2O. And then transurethral fulguration is performed on the Hunner lesion.
  Arms: TUF+HD

SUMMARY:
This study is a randomized controlled trial. Subject population is adult patients with Hunner-type interstitial cystitis. The objective of this study is to compare the therapeutic effect between the two surgical modality; TUF (transurethral fulguration of the Hunner lesion) versus TUF+HD(addition of bladder hydrodistension prior to transurethral fulguration of the Hunner lesion).

DETAILED DESCRIPTION:
Subject patients are randomly allocated to 1:1 ratio using Permuted block randomization. For TUF group, only fulguration on the Hunner lesion is performed. For TUF+HD group hydrodistension is performed for 8 minutes at pressure of 80cmH2O, and then fulguration on the Hunner lesion is performed. Therapeutic effect is evaluated using Visual Analogue Scale (VAS) pain score, O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q), Pelvic pain urgency/frequency patient symptom scale (PUF), frequency volume chart parameters, EQ-5D Health Questionnaire, Brief Pain Inventory-short form (BPI-sf), Patient Global Assessment (PGA) at the point of 1, 2, 4 and 6 months after operation. During the observational period, subject patients are not provided with any additional medical, physical or surgical treatment for symptom relief. Subject patient who complains of symptom requiring medical, physical or surgical intervention during the study period, is dropped from the study. Comparison of therapeutic efficacy between the two groups is performed using independent two sample t-test.

ELIGIBILITY:
Inclusion Criteria:

* 1. cystoscopically proven Hunner lesion, without other demonstrable lower urinary tract diseases
* 2. Adult patient aged more than 19 years
* 3. Duration of IC/BPS symptom of more than 6 months
* 4. VAS pain score more than point 4 (including point 4)
* 5. The total score of O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) symptom and problem is more than 12 with the score of pain item is more than 2
* 6. The total score of Pelvic pain urgency/frequency patient symptom scale more than point 13

Exclusion Criteria:

* 1. Patient with history of bladder hydrodistension or transurethral fulguration within the period of 3 months
* 2. Women patients who are likely to become pregnant
* 3. Patients with average voided volume more than 400ml
* 4. Patients with hematuria suspicious of malignancy
* 5. Patients with microbiologically proven urinary tract infection during the screening period
* 6. Patients with microbiologically proven recurrent urinary tract infection, more than twice during the last 6 months or more than three times of infection during the last year
* 7. Patients with previous history of genitourinary tuberculosis
* 8. Patients with previous history of genitourinary malignancy
* 9. Patients with previous history of bladder augmentation
* 10. Patient with following surgery within recent 6 months at screening; hysterectomy, midureteral or suburethral sling operation, transvaginal operation, pelvic organ prolapse surgery, vaginal delivery, Caesarean section, prostate surgery, and any other treatment that might affect bladder sensation and bladder function.
* 11. Patients with neurological diseases which might affect bladder function
* 12. patients who rely on assisted emptying ; like clean intermittent catheterization or indwelling catheterization
* 13. patients who are planning to rehabilitation treatment affect the bladder function, like intravesical electronic stimulation
* 14. patient with alcohol or drug addiction
* 15. any patient who are not fit for the study based on the investigator's decision

Ages: 29 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
inter-group difference of VAS pain score at postoperative one month | at postoperative one month
  Primary end-point is inter-group difference of VAS pain score at postoperative one month. Analysis is performed based on independent two sample t-test. ; About the VAS pain score -'VAS' is abbreviation of 'Visual Analogue Scale'. For evaluation of pain, we use 'Visual Analogue Scale' which has a range from 0 to 10 points.
  The score increases depending on the severity of the pain symptoms.

SECONDARY OUTCOMES:
inter-group differences in drop-out rate at postoperative 6 months | at postoperative 6 months
  Assessment of Drop-out rate is performed at the point of postoperative 6 months (both using the Intention-To-Treat and Per-Protocol analysis)
inter-group differences in O'Leary-Sant Interstitial Cystitis-Questionnaires | at postoperative 1 month
  O'Leary-Sant questionnaire assesses severity of symptoms on the bladder pain, frequency, urgency, nocturia, composed of symptom index and problem index
inter-group differences in O'Leary-Sant Interstitial Cystitis-Questionnaires | at postoperative 2 months
  O'Leary-Sant questionnaire assesses severity of symptoms on the bladder pain, frequency, urgency, nocturia, composed of symptom index and problem index
inter-group differences in O'Leary-Sant Interstitial Cystitis-Questionnaires | at postoperative 4 months
  O'Leary-Sant questionnaire assesses severity of symptoms on the bladder pain, frequency, urgency, nocturia, composed of symptom index and problem index
inter-group differences in O'Leary-Sant Interstitial Cystitis-Questionnaires | at postoperative 6 months
  O'Leary-Sant questionnaire assesses severity of symptoms on the bladder pain, frequency, urgency, nocturia, composed of symptom index and problem index
inter-group differences in PUF(Pelvic pain and Urgency/Frequency patient symptom scale) | at postoperative 1 month
  PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is questionnaire which evaluates symptoms of pain, urgency, and frequency and how much they bother the patient. PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is composed of two compartment; symptom score (7 items) and bother score (4 items). The symptom scores range from 2~23 points and the symptom scores range from 0~12 points. The higher the score, the worse the symptoms.
inter-group differences in PUF(Pelvic pain and Urgency/Frequency patient symptom scale) | at postoperative 2 months
  PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is questionnaire which evaluates symptoms of pain, urgency, and frequency and how much they bother the patient. PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is composed of two compartment; symptom score (7 items) and bother score (4 items). The symptom scores range from 2~23 points and the symptom scores range from 0~12 points. The higher the score, the worse the symptoms.
inter-group differences in PUF(Pelvic pain and Urgency/Frequency patient symptom scale) | at postoperative 4 months
  PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is questionnaire which evaluates symptoms of pain, urgency, and frequency and how much they bother the patient. PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is composed of two compartment; symptom score (7 items) and bother score (4 items). The symptom scores range from 2~23 points and the symptom scores range from 0~12 points. The higher the score, the worse the symptoms.
inter-group differences in PUF(Pelvic pain and Urgency/Frequency patient symptom scale) | at postoperative 6 months
  PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is questionnaire which evaluates symptoms of pain, urgency, and frequency and how much they bother the patient. PUF (Pelvic pain and Urgency/Frequency patient symptom scale) is composed of two compartment; symptom score (7 items) and bother score (4 items). The symptom scores range from 2~23 points and the symptom scores range from 0~12 points. The higher the score, the worse the symptoms.
inter-group differences in EQ-5D Health Questionnaire | at postoperative 1 month
  The EQ-5D questionnaire is a tool for brief evaluation of subject's health status. The EQ-5D questionnaire has five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has three-level; having no problems, having some or moderate problems, being unable to do/having extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number. The 5-digit number is finally converted to a single summary index by a specific formula.
inter-group differences in EQ-5D Health Questionnaire | at postoperative 2 months
  The EQ-5D questionnaire is a tool for brief evaluation of subject's health status. The EQ-5D questionnaire has five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has three-level; having no problems, having some or moderate problems, being unable to do/having extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number. The 5-digit number is finally converted to a single summary index by a specific formula.
inter-group differences in EQ-5D Health Questionnaire | at postoperative 4 months
  The EQ-5D questionnaire is a tool for brief evaluation of subject's health status. The EQ-5D questionnaire has five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has three-level; having no problems, having some or moderate problems, being unable to do/having extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number. The 5-digit number is finally converted to a single summary index by a specific formula.
inter-group differences in EQ-5D Health Questionnaire | at postoperative 6 months
  The EQ-5D questionnaire is a tool for brief evaluation of subject's health status. The EQ-5D questionnaire has five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has three-level; having no problems, having some or moderate problems, being unable to do/having extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number. The 5-digit number is finally converted to a single summary index by a specific formula.
Brief Pain Inventory-short form (BPI-sf) | at postoperative 1 month
  Brief Pain Inventory-short form (BPI-sf) is composed of two domains measured by the "pain severity" and the "pain interference", Pain severity compartment is composed of 4 items, and pain interference compartment is composed of 7 items (of 24-hour recall period). Each item has 0-10 scales. Brief pain severity score is calculated by adding the scores of 4 questions and then dividing by 4. Brief pain interference score is calculated by adding the scores for 7 questions and then dividing by 7.
Brief Pain Inventory-short form (BPI-sf) | at postoperative 2 months
  Brief Pain Inventory-short form (BPI-sf) is composed of two domains measured by the "pain severity" and the "pain interference", Pain severity compartment is composed of 4 items, and pain interference compartment is composed of 7 items (of 24-hour recall period). Each item has 0-10 scales. Brief pain severity score is calculated by adding the scores of 4 questions and then dividing by 4. Brief pain interference score is calculated by adding the scores for 7 questions and then dividing by 7.
Brief Pain Inventory-short form (BPI-sf) | at postoperative 4 months
  Brief Pain Inventory-short form (BPI-sf) is composed of two domains measured by the "pain severity" and the "pain interference", Pain severity compartment is composed of 4 items, and pain interference compartment is composed of 7 items (of 24-hour recall period). Each item has 0-10 scales. Brief pain severity score is calculated by adding the scores of 4 questions and then dividing by 4. Brief pain interference score is calculated by adding the scores for 7 questions and then dividing by 7.
Brief Pain Inventory-short form (BPI-sf) | at postoperative 6 months
  Brief Pain Inventory-short form (BPI-sf) is composed of two domains measured by the "pain severity" and the "pain interference", Pain severity compartment is composed of 4 items, and pain interference compartment is composed of 7 items (of 24-hour recall period). Each item has 0-10 scales. Brief pain severity score is calculated by adding the scores of 4 questions and then dividing by 4. Brief pain interference score is calculated by adding the scores for 7 questions and then dividing by 7.
Patient Global Assessment (PGA) | at postoperative 1 month
  Patient Global Assessment (PGA) is composed of a single questionnaire assessing the subjective patients-reported outcome. The question is "How is your bladder condition today?". The patients choose one of the following five answers; very-good, god, moderate, bad, very bad.
Patient Global Assessment (PGA) | at postoperative 2 months
  Patient Global Assessment (PGA) is composed of a single questionnaire assessing the subjective patients-reported outcome. The question is "How is your bladder condition today?". The patients choose one of the following five answers; very-good, god, moderate, bad, very bad.
Patient Global Assessment (PGA) | at postoperative 4 months
  Patient Global Assessment (PGA) is composed of a single questionnaire assessing the subjective patients-reported outcome. The question is "How is your bladder condition today?". The patients choose one of the following five answers; very-good, god, moderate, bad, very bad.
Patient Global Assessment (PGA) | at postoperative 6 months
  Patient Global Assessment (PGA) is composed of a single questionnaire assessing the subjective patients-reported outcome. The question is "How is your bladder condition today?". The patients choose one of the following five answers; very-good, god, moderate, bad, very bad.
frequency volume chart parameters | at postoperative 1 month
  frequency volume chart is a tool for assessment of micturition time, volume of urination and urgency episode. 24-hr frequency of micturition, maximum voided volume, episode of urgency, and nocturia is evaluated.
frequency volume chart parameters | at postoperative 2 months
  frequency volume chart is a tool for assessment of micturition time, volume of urination and urgency episode. 24-hr frequency of micturition, maximum voided volume, episode of urgency, and nocturia is evaluated.
frequency volume chart parameters | at postoperative 4 months
  frequency volume chart is a tool for assessment of micturition time, volume of urination and urgency episode. 24-hr frequency of micturition, maximum voided volume, episode of urgency, and nocturia is evaluated.
frequency volume chart parameters | at postoperative 6 months
  frequency volume chart is a tool for assessment of micturition time, volume of urination and urgency episode. 24-hr frequency of micturition, maximum voided volume, episode of urgency, and nocturia is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology and Urological Science Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Currently, we do not plan to share patient data with third parties.

REFERENCES:
- [Background] Malde S, Palmisani S, Al-Kaisy A, Sahai A. Guideline of guidelines: bladder pain syndrome. BJU Int. 2018 Nov;122(5):729-743. doi: 10.1111/bju.14399. Epub 2018 Jun 13. PMID 29777618
- [Background] Kirk PS, Santiago-Lastra Y, Qin Y, Stoffel JT, Clemens JQ, Cameron AP. The effects of cystoscopy and hydrodistention on symptoms and bladder capacity in interstitial cystitis/bladder pain syndrome. Neurourol Urodyn. 2018 Aug;37(6):2002-2007. doi: 10.1002/nau.23555. Epub 2018 Mar 22. PMID 29566264
- [Background] Bosch PC. A Randomized, Double-blind, Placebo-controlled Trial of Certolizumab Pegol in Women with Refractory Interstitial Cystitis/Bladder Pain Syndrome. Eur Urol. 2018 Nov;74(5):623-630. doi: 10.1016/j.eururo.2018.07.026. Epub 2018 Jul 30. PMID 30072210
- [Background] Akiyama Y, Niimi A, Nomiya A, Yamada Y, Nakagawa T, Fujimura T, Fukuhara H, Kume H, Igawa Y, Homma Y. Extent of Hunner lesions: The relationships with symptom severity and clinical parameters in Hunner type interstitial cystitis patients. Neurourol Urodyn. 2018 Apr;37(4):1441-1447. doi: 10.1002/nau.23467. Epub 2018 Jan 9. PMID 29315774
- [Derived] Son HS, Yoon H, Lee HS, Kim JH. Prospective randomized controlled trial comparing fulguration versus fulguration and hydrodistension for Hunner-type interstitial cystitis/bladder pain syndrome. World J Urol. 2022 Aug;40(8):2071-2076. doi: 10.1007/s00345-022-04062-8. Epub 2022 Jun 15. PMID 35704106